CLINICAL TRIAL: NCT00174096
Title: The Role of Stromal Cell-Derived Factor-1 (SDF-1)/CXC Chemokine Receptor 4 (CXCR4) in Metastasis of Laryngeal and Hypopharyngeal Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700624
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2006-03-31 (Estimated); Status verified 2005-06

CONDITIONS: Laryngeal Cancer; Hypopharyngeal Cancer; Metastasis
Keywords: laryngeal cancer; hypopharyngeal cancer; CXCR4; stromal-cell-derived factor-1(SDF-1); metastasis
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to investigate the relationship between SDF-1/CXCR4 and metastasis of laryngeal and hypopharyngeal squamous cell carcinomas.

DETAILED DESCRIPTION:
Cancer of the larynx and hypopharynx remains the third most common head and neck malignancy, constituting about 20% of all tumors. Squamous cell carcinoma (SCC) is the most common histopathologic type of the laryngeal and hypopharyngeal malignancies, accounting for more than 90% of cancers occurring in this region. Lymph node metastasis directly affects the prognosis of patients with laryngeal and hypopharyngeal SCC. The presence of lymph node metastasis significantly reduces the probability of regional control and survival. Furthermore, the American Cancer Society shows no trend toward an improvement in 5-year survival rates between patients diagnosed in 1974 to 1976 and 1989 to 1995.

Tumor metastasis is the hallmark of malignancy, and is probably a result of the interaction between tumor cells and a supportive microenvironment. Malignant cells that have the capability to metastasize to a particular organ may have various properties supporting their tissue invasion or growth such as enhanced adherence to the microvascular cells of the organ, higher responsiveness to chemotactic signals released from the target organs and increased response to local soluble or tissue associated growth signals in the target organ. Though several molecules expressed or produced in cancer cells are considered the metastatic factors, it remains unknown which factors produced by the lymph node or tissue affect the metastasis of cancer cells.

Chemokines are a large family of pro-inflammatory polypeptide cytokines, consisting of small (7-15 kDa), structurally related heparin-binding proteins. They are grouped into CXC chemokines and CC chemokines, on the basis of the characteristic presence of four conserved cysteine residues. Chemokines are produced locally in the tissues and act on target cells through G-protein-coupled receptors, which are characterized structurally by seven transmembrane spanning domains. Chemokines are involved in the attraction and activation of mononuclear and polymorphonuclear leukocytes to sites of inflammatory responses, bacterial or viral infections, allergy, cardiovascular diseases and wound healing. Chemokines are known to also function as regulatory molecules in the leukocyte maturation, trafficking, and homing of T and B lymphocytes, in the development of lymphoid tissues, and in dendritic cell maturation. Other functions of chemokines have been described more recently, particularly for the CXC chemokines. The role of chemokines in malignant tumors is not clear yet. Some chemokines may enhance innate or specific host immunity against tumor dissemination. On the other hand, some may advocate tumor growth and metastasis by promoting tumor cell proliferation, migration or angiogenesis in tumor tissue. Reports have suggested that several types of cancer, such as breast, ovary, prostate, kidney, brain, lung, and thyroid, expressed the chemokine receptor and used the chemokines to metastasize to the target organ as in the homing of hematopoietic cells.

SDF-1 belongs to the CXC chemokine family and is a ligand for CXCR4. SDF-1 was initially cloned by Tashiro et al. and later identified as a growth factor for B cell progenitors, a chemotactic factor for T cells and monocytes, and in B-cell lymphopoiesis and bone marrow myelopoiesis. Most of the chemokine receptors interact with pleural ligands, and vice versa, but the SDF-1/CXCR4 receptor ligand system has been shown to involve a one-on-one interaction. Recently, several studies have been conducted to detect the mRNA expression of CXCR4 and SDF-1 in solid tumors. The results are not uniform, and the relevance to cancer progression is not determined. Sehgal et al. concluded that CXCR4 plays an important role of proliferation and tumorigenic properties of human glioblastoma tumors. Muller et al. have reported that SDF-1 signaling through CXCR4 interaction appears to determine the directional migration of breast cancer cells through the basement membrane. Furthermore in vivo, the interaction between SDF-1 and CXCR4 significantly represses the metastatic potential of breast cancer cells to lymph node and lung. Barnard and his colleagues showed the contrary results that CXCR4 mRNA expression was reduced in hepatocellular carcinoma tissue when compared with noncancerous tissue, but was not changed in colon, esophageal, and gastric cancer. They also found reduced mRNA expression of SDF-1 in these malignant tissues. Thus, there is a diversity of views on the role of the SDF-1/CXCR4 receptor ligand system in malignant tissues. And such studies are limited in laryngeal and hypopharyngeal cancer.

Metastasis of laryngeal and hypopharyngeal cancer occurs frequently through the lymphatic system, and metastasis is a key prognostic factor for the disease. Evaluation of the relationship between SDF-1/CXCR4 system and metastasis in laryngeal and hypopharyngeal cancer could help us understand whether this system is important in the metastasis of this disease.

We hypothesized that SDF-1/CXCR4 (ligand/receptor) system plays an important role in laryngeal and hypopharyngeal cancer metastasis. To test this hypothesis, we will investigate:

1. the distribution of CXCR4 protein expression in cancer and lymph node tissues by means of immunohistochemical analysis of tissue samples obtained from surgical operation
2. the relationship between CXCR4 expression and clinicopathological findings with special reference to cancer metastasis
3. the expression of SDF-1 and CXCR4 in the cancer cell line cells and tissues
4. the chemotactic activity and the growth-promoting effect of SDF-1 on cancer cell line cells
5. the role of Src, MAPK, and Akt signal transduction pathway in this response
6. the effect of the blocking agent on this response.

Undoubtedly, the findings of this study will help us understand whether SDF-1/CXCR4 system could be a focal point of anti-cancer research. If laryngeal and hypopharyngeal SCC that express high levels of CXCR4 show a consistently higher incidence of lymphatic and distant metastasis, then blocking SDF-1/CXCR4 signaling may be a novel approach to inhibit metastasis in these patients. The development of SDF-1/CXCR4 system antagonists will provide an opportunity to improve the survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Laryngeal or hypopharyngeal squamous cell carcinoma

Exclusion Criteria:

* Pathology other than SCC

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Ting Tan, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan